CLINICAL TRIAL: NCT06054906
Title: Neoadjuvant of Sintilimab Combined Weekly Metronomic Chemotherapy (PLOF) for Resectable Locally Advanced Gastric Cancer : a Phase Il Study
Brief Title: Neoadjuvant of Sintilimab Combined Weekly Metronomic Chemotherapy (PLOF) for Resectable Locally Advanced Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhongguang Luo, MD, Chief Physician, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2022-1018
Record Dates: First submitted 2023-09-12; First posted 2023-09-26 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- sintilimab+metronomic PLOF (Experimental): sintilimab therapy(200mg, iv,d1,Q3W, 2cycles)and PLOF chemotherapy (Paclitaxel 60 mg/m2, oxaliplatin 50 mg/m2, 5-fluorouracil 425mg/m2, d1, QW, 6cycles) followed by adjuvant sintilimab therapy(200mg, iv,d1,Q3W, 2cycles)and PLOF chemotherapy (Paclitaxel 60 mg/m2, oxaliplatin 50 mg/m2, 5-fluorouracil 425mg/m2, d1, QW, 6cycles) neoadjuvant chemotherapy (8 weeks) preceding surgery (3 weeks after completion of chemotherapy) followed by adjuvant chemotherapy (16 weeks, begin within 12 weeks after surgery)
  Interventions: Drug: sintilimab+metronomic PLOF

INTERVENTIONS:
Drug: sintilimab+metronomic PLOF — Drug: Sintilimab 200mg iv d1 Q3W, 2cycles
  Drug: Paclitaxel 60 mg/m2, d1, QW,6cycles
  Drug: Oxaliplatin 50 mg/m2, d1, QW, 6cycles
  Drug: 5-fluorouracil 425mg/m2 ,d1 ,QW, 6cycles

SUMMARY:
To evaluate efficacy and safety of Neoadjuvant of Sintilimab Combined Weekly Metronomic Chemotherapy (PLOF) in resectable locally advanced gastric cancer.

DETAILED DESCRIPTION:
This is a single-arm clinical study to enroll 50 patients with gastric cancer (cTNM diagnosis of cT3-4aN1-3M0). Each enrolled patient will be assigned a case number. Both this case number and the patient's initials will be entered on each page of the case report form.

Enrolled patients receive a neoadjuvant regimen of POLF in combination with sindilizumab: preoperatively, they receive a POLF regimen (paclitaxel 60 mg/m2, oxaliplatin 50 mg/m2, and 5-fluorouracil 425 mg/m2) administered once weekly for a total of 6 doses, and in combination with sindilizumab 200 mg intravenously once every 3 weeks for a total of 2 doses. Upon completion of the evaluation, patients whose tumors were judged to be resectable underwent radical surgery and received six postoperative doses of the POLF regimen and two doses of Sindilizumab as adjuvant therapy.

Postoperative imaging evaluations will be performed every three months until disease recurrence. Survival follow-up was performed every three months after disease recurrence. Patients will receive neoadjuvant therapy for 6 weeks preoperatively and adjuvant therapy for 6 weeks postoperatively unless intolerable toxicity occurs, the patient refuses to continue treatment, or treatment is delayed beyond 3 weeks. Patients will be under study observation during treatment and 30 days after treatment termination, and will receive long-term follow-up for 5 years postoperatively. Ultimately, pCR and MPR will be the primary study endpoints, and ORR, DCR, 2-year PFS rate, 3-year OS rate and safety will be the secondary study endpoints to evaluate the efficacy and safety of the neoadjuvant regimen of POLF combined with sindilizumab, as well as to explore the immune activation effect and mechanism of the regimen using peripheral blood and tumor tissue samples.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written Informed Consent Form
2. Male or female, age ≥ 18 years old
3. Histologically confirmed gastric adenocarcinoma, diagnosed as locally progressive according to the AJCC 8th ed, cTNM diagnosis of cT3-4aN1-3M0 and resectable lesion as assessed by the investigator
4. No prior systemic therapy such as surgery, radiotherapy, or immunotherapy for the disease at hand
5. Consent to radical surgical treatment and no contraindications to surgery as determined by the surgeon
6. ECOG PS: 0-1 score
7. Expected survival > 6 months
8. Adequate organ function, must meet the following laboratory specifications:

   8.1 Absolute neutrophil count (ANC) ≥ 1.0x10^9/L; 8.2 Platelets ≥ 80x10^9/L; 8.3 Hemoglobin > 7g/dL; 8.4 Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (Total bilirubin > 1.5 x ULN but direct bilirubin ≤ ULN are allowed to be enrolled); 8.5 AST, ALT ≤ 2.5×ULN; 8.6 Blood creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 60 ml/min; 8.7 INR or PT ≤ 1.5 times ULN; 8.8 TSH within normal range (Enrollment allowed if baseline TSH is outside normal range but FT4 is within normal range); 8.9 Myocardial enzyme profile within normal range;
9. Negative pregnancy test in women of childbearing age
10. Need to use contraception with an annual failure rate of less than 1% if there is a risk of conception

Exclusion Criteria:

1. Endoscopically show signs of active bleeding from the lesion
2. Current participation in an interventional clinical study or treatment with another investigational drug or use of an investigational device within 4 weeks prior to the first dose of study drug
3. Prior therapy with anti-PD-1, anti-PD-L1, or anti-PD-L2 agents, or agents targeting CTLA-4, OX-40, CD137, etc.
4. Diagnosis of a malignant disease other than gastric cancer within 5 years prior to the first dose of therapy
5. Active autoimmune disease requiring systemic therapy within 2 years prior to the first dose of the drug
6. Live vaccination within 30 days prior to the first administration of the drug
7. Have received systemic systemic therapy with proprietary Chinese medicines with antitumor indications or immunomodulatory drugs within 2 weeks prior to the first administration of the drug
8. Have received systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of treatment
9. Has not fully recovered from any intervention-induced toxicity and/or complications (excluding malaise or alopecia) prior to initiation of therapy
10. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation
11. Known hypersensitivity to drugs used in this study
12. Known history of HIV infection
13. Untreated active hepatitis B
14. Active HCV infection
15. Pregnant or lactating women
16. The presence of any serious or uncontrolled systemic disease
17. Other factors that, in the judgment of the investigator, may affect the outcome of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with no residual surviving tumor cells in resection specimens and lymph nodes | up to 6 weeks after first dosing
  Pathological complete response rate (pCR), defined as the proportion of participants with no residual viable tumor cells on microscopy and negative lymph nodes as a percentage of all participants. We will evaluate pathological complete response rate of primary tumor and locally metastatic lymph nodes after 6 weeks of neoadjuvant therapy.
Percentage of participants with ≤10% tumor cell survival in resection specimens | up to 6 weeks after first dosing
  Major pathologic response (MPR) rate, defined as the proportion of participants with ≤10% surviving tumor cells in the resection specimen as a percentage of all participants. We will evaluate major pathological response rate of primary tumor and locally metastatic lymph nodes after 6 weeks of neoadjuvant therapy.

SECONDARY OUTCOMES:
Percentage of participants achieving complete remission (CR) and partial remission (PR) after treatment | 2 to 6weeks after the end of treatment
  Objective remission rate (ORR), the percentage of participants whose tumors shrink by a certain amount and remain there for a certain period of time, including complete remission (CR) and partial remission (PR). CR (Complete remission): Complete disappearance of the target lesion, with no new lesions produced, and lasting for more than 4 weeks. PR (Partial remission): the sum of the largest diameters of the target lesions is reduced by more than 30%, and lasts for more than 4 weeks.
Percentage of participants achieving remission (PR+CR) and lesion stabilization (SD) after treatment | 2 to 6weeks after the end of treatment
  Disease control rate (DCR) is the percentage of participants who achieve remission (PR+CR) and stabilization of lesions (SD) after the treatment. Stable disease (SD) means that the sum of the largest diameters of the tumor lesions has not shrunk to PR, or has not enlarged to PD.
2-year progression-free survival (PFS) rate | From enrollment to study completion, assessed up to 2 years
  Percentage of participants who survived or were free of tumor progression from enrollment to the second year of follow-up.
3-year overall-survival (OS) rate | From enrollment to study completion, assessed up to 3 years
  Percentage of participants who survived from enrollment to the third year of follow-up.
Number of participants with treatment-related adverse events as assessed by NCI-CTC | From enrollment to study completion, assessed up to 3 years
  Toxicity deaths and early withdrawal from treatment due to toxic effects will be described. Toxicity assessment of adverse events and serious adverse events (SAEs) using the NCI-CTC.

OTHER OUTCOMES:
Number of immune cells in peripheral blood | From enrollment to study completion, assessed up to 3 years
  Peripheral blood will be analyzed for the number of immune cells after applying flow cytometry and mRNA sequencing.
Proportion of immune cells in peripheral blood | From enrollment to study completion, assessed up to 3 years
  Peripheral blood will be analyzed for the proportion of immune cells after applying flow cytometry and mRNA sequencing.
Number of immune cells in tumor tissues | From enrollment to study completion, assessed up to 3 years
  Apply mRNA sequencing, immunohistochemistry and immunofluorescence to analyze the number of immune cells in tumor tissues, including CTL, Treg, DC, TAM, MDSC, NK, NKT and so on.
Distribution of immune cells in tumor tissue | From enrollment to study completion, assessed up to 3 years
  Apply mRNA sequencing, immunohistochemistry and immunofluorescence to analyze the distribution of immune cells in tumor tissues, including CTL, Treg, DC, TAM, MDSC, NK, NKT and so on.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No